CLINICAL TRIAL: NCT05225129
Title: Effects Of Blood Flow Restriction Exercise Applications On Physical Fitness Parameters and Sporting Motivation in Canoe Athletes
Brief Title: Effects Of Blood Flow Restriction Exercise Applications On Physical Fitness Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Burçin Uğur Tosun, Principal Investigator, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/12/31
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Physical Performance
Keywords: blood flow restriction; physical parameters; sporting motivation; canoe
MeSH Terms: interventions — Blood Flow Restriction Therapy; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): Resistance training will be applied to the training group, equivalent to 30% of 1 maximum repetition with blood flow restricted exercise for 8 weeks , 2 days in a week.
  Interventions: Other: blood flow restriction exercise
- Control Group (No Intervention): Resistance training will be applied to the control group, equivalent to 30% of 1 maximum repetition without blood flow restriction for 8 weeks , 2 days in a week.

INTERVENTIONS:
Other: blood flow restriction exercise — blood flow restricted exercise, resistance training will be applied, corresponding to 30% of 1 maximum repetition for 8 weeks, 2 days in a week
  Other Names: resistance exercise
  Arms: Training Group

SUMMARY:
Aim: The aim of the study; during the non-race season, blood flow-restricted exercises applied in addition to routine training programs to determine the effects on physical fitness parameters and sportive motivation of male canoe athletes aged 18 and over and to compare the results between the groups.

Method: Male athletes aged 18 and over who are licensed and actively engaged in canoeing in Turkey will be included in the study. Subjects will be divided into two groups , training and control. The training group will be given blood flow restricted exercise for 8 weeks and resistance training equivalent to 30% of 1 maximum repetition. In the control group, 30% of 1 MT of resistance training will be applied for 8 weeks without blood flow restriction. Before and after, athletes will be evaluated with sport-specific performance tests, muscle thickness measurement with ultrasound, isokinetic measurement of hamstring and quadriceps muscles at a speed of 60°/sec and 300°/sec. In addition, the muscles of the athletes will be evaluated with dynamic muscular measurements.

DETAILED DESCRIPTION:
The first evaluation will be made before the 8-week training, and the second evaluation will be made at the end of the 8-week training. Both groups will be re-evaluated for follow-up at 6 and 12 months from the start of the study. In the 4th week, it is aimed to improve the exercise protocols by increasing the number of sets and repetitions in both groups.

The training will start with a 10-minute warm-up exercise on the static bike, and then stretching exercises will be applied. The athlete is dressed in the KAK apparatus and the pressure is given continuously so that it is on the device. In the 30-minute CAC exercise training, the athlete will complete the resistance exercises on the Leg Press, Leg Curl, Leg Calf Raise, Quadriceps Extension machines while attached to the device.

In the exercise prescription, which is planned as 3 sets of 10 repetitions, a rest period of 60 seconds will be given between sets. A 10-minute cool-down period will be added at the end of the training.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Being a licensed athlete for at least 2 years,
* No history of orthopedic injury in the last 6 months
* Athletes who have been doing resistance exercise for at least 5 years

Exclusion Criteria:

* Presence of disease that will cause endothelial dysfunction (hypertension, cardiovascular diseases, neurological diseases, atherosclerosis)
* History of deep vein thrombosis and peripheral vascular disease
* Presence of acute infection
* Cancer cases
* Having undergone a surgical operation due to trauma in the last 6 months

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-10-22 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Changes in the sportive performance will be measured by ergometer | At the beginning and at the end of 8 weeks
  Indoor ergometer will be used to determine the sportive performance changes of canoe athletes.
Changes in muscle thickness will be measured by ultrasound | At the beginning and at the end of 8 weeks
  The thickness measurements of the Rectus Femoris, Vastus Medialis Obliqus, Vastus Lateralis and Hamstring muscles and the area measurements of the rectus femoris and hamstring muscles will be measured by the sports physician.
Quadriceps and Hamstring muscle strength, endurance, Ham/Quad ratio will be evaluated with an isokinetic dynamometer. | At the beginning and at the end of 8 weeks
  Angular velocities; 60 degrees/sec, 300 degrees/sec will be measured bilaterally with the Biodex System 3. For 60 degrees / sec, the athlete will do 5 repetitions, and for 300 degrees / sec, the athlete will do 15-20 repetitions. Before both measurements, evaluation will begin after 3 rewarmings.
In the Dynamic Measurement of Muscular Strength, a repetitive maximum method is used to measure the force with the dynamic method. | At the beginning and at the end of 8 weeks
  It is performed with an appropriate starting weight close to but below the person's maximal lifting capacity for any muscle group. After the first repetition, the weight is lifted until the maximum lifting force is reached. It determines the maximum weight that athletes can lift at once in normal joint movement.

CONTACTS AND LOCATIONS:
Overall Officials: Berkiye Kırmızıgil, Asst. Prof., Study Chair — Eastern Mediterranean University
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No